CLINICAL TRIAL: NCT04740411
Title: An Online Wellness Intervention for American College Students: Investigating the Efficacy of The Common Elements Toolbox
Brief Title: Online Wellness Intervention for College Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pennsylvania (Other)
Collaborators: Indiana University (Other); Ohio State University (Other); University of Missouri, St. Louis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 844589
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Depression; Anxiety; Well-being
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Common Elements Toolbox (COMET) (Experimental)
  Interventions: Behavioral: The Common Elements Toolbox (COMET)
- Wait-list control condition (No Intervention)

INTERVENTIONS:
Behavioral: The Common Elements Toolbox (COMET) — COMET is an online unguided self-help intervention that lasts approximately 60-80 minutes.
  Arms: Common Elements Toolbox (COMET)

SUMMARY:
We are evaluating the effects of an online single-session mental health intervention (the Common Elements Toolbox; COMET). To evaluate COMET, we are conducting a randomized controlled trial with college students attending American universities. Students will be randomized to the COMET condition or to a wait-list control condition.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old and a student at a participating university. Access to the internet.

Exclusion Criteria:

* Cannot have participated in a previous version of COMET.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Patient Health Questionnaire-9 (PHQ-9) | Up to 8 weeks post-intervention
  Depression questionnaire. Scores range from 0 to 27. Lower scores indicate less depression.
Change in the Generalized Anxiety Disorder Screener-7 (GAD-7) | Up to 8 weeks post-intervention
  Anxiety questionnaire. Total scores range from 0-21. Lower scores indicate less anxiety.
Change in the Short Warwick-Edinburgh Mental Well-being Scale | Up to 8 weeks post-intervention
  Subjective Well-being questionnaire. Total scores range from 7 to 35. Higher values indicate higher well-being scores.
Change in items from the PERMA Profiler (positive emotion and negative emotion subscales). | Up to 8 weeks post-intervention
  Well-being questionnaire with questions related to positive emotion, engagement, relationships, meaning, accomplishment, negative emotion, and health. Scores on each item range from 0 to 5. Lower scores indicate less well-being. We are using a shortened version of this questionnaire with 12 items. We have also modified the items to ask participants about their experiences over the past 48 hours. We predict that our intervention will produce changes in the positive emotion and negative emotion subscales. Each subscale consists of 3 items.

SECONDARY OUTCOMES:
Ratings on the Acceptability of Intervention Measure (AIM) | Immediately after the intervention
  Questionnaire measuring the acceptability of an intervention. Acceptability refers to the perception that a given treatment is agreeable or satisfactory. The total score ranges from 4 to 20. Higher scores indicate higher acceptability ratings.
Ability to Cope with COVID-19 | Up to 8 weeks post-intervention
  2 questions related to their ability to cope with stressors over the past two weeks relating to the COVID-19 pandemic. Participants answered these questions on a 7-point Likert Scale, from "strongly disagree" to "strongly agree". Specifically, we asked participants: a) if they have been able to handle lifestyle changes due to the coronavirus and b) if the pandemic has had an extremely negative impact on their life.
Change in Secondary Control | Up to 8 weeks post-intervention
  We administered three items to assess secondary control, derived from the Secondary Control Scale for Children (Weisz et al., 2010). The items are scored on a 4-point Likert scale, ranging from 0 ("Very false") to 3 ("Very true"). Scores on each item range from 0-4, with higher scores indicating more secondary control.
Change in the Positive and Negative Affect Schedule | Up to 8 weeks post-intervention
  Questionnaire measuring positive affect and negative affect. Scores on the positive affect subscale range from 10-50, with higher scores representing higher levels of positive affect. Scores on the negative affect subscale range from 10-50, with lower scores representing lower levels of negative affect.
Perceived Utility Ratings | Immediately after the intervention
  Participants were asked to rate three items relating to the perceived utility of each module. Specifically, we asked participants: How helpful the module was How engaging the module was How much they will continue applying content from the module. Higher scores indicate greater perceived utility.
Change in the Perceived Stress Scale-4 | Up to 8 weeks post-intervention
  Questionnaire measuring perceived stress. Scores range from 0-16, with higher scores indicating greater stress.
Change in the Gratitude Adjective Checklist | Up to 8 weeks post-intervention
  Gratitude measure. Three items rated on a 1-5 scale with total scores ranging from 3-15. Higher scores indicate higher levels of gratitude.
Change in the Self-kindness subscale of the Self-Compassion Scale | Up to 8 weeks post-intervention
  Self-compassion measure. We are using the 5-item self-kindness subscale. Participants will provide values ranging from 1 to 5. These values will be summed to create a total score on this scale ranging from 5 to 25, with higher scores representing higher levels of self-compassion.
Change in Cognitive Restructuring | Up to 8 weeks post-intervention
  We administered three items to assess cognitive restructuring, derived from the cognitive reappraisal subscale of the Emotion Regulation Questionnaire. Scores range from 3-21, with higher scores representing a higher amount of cognitive restructuring.
Change in items from the Behavioral Activation for Depression Scale | Up to 8 weeks post-intervention
  Behavioral Activation Measure. We selected 3 items from the BADS to use to assess changes in behavioral activation. The scores for these three items are summed to give a total score from 0-18. Higher scores represent higher levels of behavioral activation.
Beck Hopelessness Scale | Up to 8 weeks post-intervention
  Hopelessness Questionnaire. Total score ranges from 0 to 4. Higher scores indicate less hope (more hopelessness).
Change in module-specific skills | Up to 8 weeks post-intervention
  We are administering 4 items designed to detect cognitive or behavioral changes that relate to each intervention module.
  Cognitive restructuring: "Over the past two weeks, I have been able to manage negative thoughts."
  Behavior activation: "Over the past two weeks, I have intentionally spent time performing hobbies and activities that make me happy."
  Gratitude: "Over the past two weeks, I have been able to focus my attention toward noticing and appreciating good things."
  Self-compassion: "Over the past two weeks, I have been able to treat myself with empathy and compassion."
  For each item, participants respond using a 7-point scale ranging from strongly disagree to strongly agree. Higher scores indicate favorable cognitions and behaviors related to each construct.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided